CLINICAL TRIAL: NCT03909919
Title: Functional Parameters Indicative of Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD. Titular Doctor Physiotherapy Department, University of Malaga. Principal investigator., University of Malaga
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Funnel study
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Kinematics; Validation; Functional task
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart Failure (Experimental): Heart Failure patients Subjects diagnosed with heart faikure, who will receive the best treatment of clinical practice, will be recruited. They must be more than 70 years old.
  Interventions: Procedure: Standard Care or Usual Clinical Practice
- Healthy Subjects (Active Comparator): Healthy Subjects/ Match control Healthy subjects of the same age as people with heart failure.
  Interventions: Procedure: Standard Care or Usual Clinical Practice

INTERVENTIONS:
Procedure: Standard Care or Usual Clinical Practice — The guidelines for the management according to the heart failure in primary care will be the treatment guidelines for the Standard Care.

SUMMARY:
The present study aims to validate the kinematic analysis obtained by two motion capture instruments for the functional objective assessment of elderly patients with Heart Failire (HF) and to develop a new functional index formed by kinematic parameters and other functional objective parameters and scales which may be impaired in patients with HF and they could allow the stratification of these patients based on different levels of functional impairment.

DETAILED DESCRIPTION:
Cardiovascular diseases carried on being the leading cause of disability due to noncommunicable diseases from 1990 to 2016. Within cardiovascular diseases, it has been estimated that heart failure (HF) has a prevalence in the population of approximately 2% to 3%. However, it is the only cardiovascular disease that is increasing in incidence and prevalence due to the aging of the world population, since the prevalence of this disease increases with age. Furthermore, heart failure represents the most important hospital diagnosis in older adults, being the main cause of hospital admissions for people older than 65 years and contributing to the increase of medical care costs.

Subjects with HF use to show a reduced aerobic capacity, a decreased muscle strength in the lower limbs, low weekly physical activity, intolerance to exercise and a lower walking speed than healthy subjects of the same age. In general, patients with heart failure have altered functional capacities and experience a decline in the ability to carry out activities of daily living and suffer a reduced quality of life. When it is assessed functional parameters in patients with heart failure, the maximum oxygen consumption (V0₂ max) obtained from a cardiopulmonary exercise test is considered the gold standard measure of cardiovascular functional capacity. Moreover, some functional tests have been used, such as the 6-Minute Walking Test, which provides an indirect measure of cardiovascular functional capacity, and the Short Physical Performance Battery (SPPB), which also provides a useful and indirect indication of muscle functional capacity. However, at the time of diagnosing or classifying patients with heart failure, the functional assessment does not use to be considered. The implementation of diagnostic guidelines or a functional assessment based on evidence can be important to improve prognosis and quality of life in patients with HF.

Therefore, there is a need to identify functional markers related to functionality that are indicative of heart failure. For this, it is necessary to use instruments to measure functional variables that must be valid and reliable, as established by the COSMIN taxonomy. Kinematic measurements allow quantifying normal and pathological movements, quantifying the degree of deterioration, planning rehabilitation strategies and evaluating the effect of various interventions. Inertial sensors and depth cameras are accurate and reliable methods for the kinematic analysis of human movement, in addition to presenting a good correlation of kinematic data between them.

Currently, it can be used the Simmer3 Inertial Sensor and 3D motion capture systems with a camera to analyse kinematics and these instruments are being integrated as a rehabilitation tool in patients. The use of Shimmer3 Inertial Sensor and 3D motion capture cameras would help to find fast and cheap assessment methods for professionals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 70 years.
* Healthy subjects and subjects diagnosed with Heart failure.
* Subjects able of filling out questionnaires and performing functional tests.
* subjects who are in a clinical stability and optimal treatment phase.

Exclusion Criteria:

* Participants with cardiac pathologies other than heart failure.
* Score in the NYHA scale equal to 4.
* Hospitalization in a period of time equal to or less than 3 months.
* Score on the Mini-Mental scale below 24.
* Inability to get up from the chair at least 5 times or 30 seconds.
* Inability to walk for 6 minutes.
* Inability to walk independently without a walking assistance device (cane, crutch or walker).
* Subjects participating in an experimental study where they receive a treatment.
* Inability to provide informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Motion parameters | 1 hour
  Kinematic parameters will be analysed using an inertial sensor included in the Shimmer3 instrument during the performance of different functional task.
Kinematic analysis by 3D motion capture | 1 hour
  A camera will perform a motion capture of the functional task. This system will calculate the displacement and the time of the functional task.
Responsiveness | 1 hour
  The Responsiveness Box of COSMIN checklist will be used to determinate the response to change of the Shimmer 3 Inertial Sensor and the 3D cameras. All possible items will be followed.
Reliability | 1 hour
  The Reliability Box of COSMIN checklist will be used to determinate the Test-Retest reliability of the Shimmer3 Inertial Sensor and the 3D cameras. All possible items will be followed.

SECONDARY OUTCOMES:
abbreviated comprehensive geriatric assessment (aCGA): a questionnaire formed by items originating from four different scales. | 15 minutes
  Questionnaire used to assess functional, emotional and cognitive components. It is composed of 15 items from the 4 instruments such as the geriatric depression scale (GDS), the Mini-Mental State Examination (MMSE), activities of daily living (ADL) using the Katz index and instrumental activities of daily living (IADL) using the Lawnton & Brody scale. The score varies from 0 to 30 points, giving 1 point to each of the items of the GDS (4 points in total), 12 to the 3 items from the scale of Lawton & Brody, 8 points to the 4 items from the MMSE and 6 points to the 3 items from the Katz index.
SARC-F | 10 minutes
  It is a simple questionnaire to rapidly diagnose Sarcopenia. It is composed by 5 components: Strength, Assistance to walk, Get up from a chair, Climb stairs and Falls. Scores range from 0 to 10, with 0 to 2 points for each component. A score equal to or greater than 4 could predict sarcopenia and poor results.
Cardiopulmonary function | 1 hour
  The heart rate will be assessed using the ECG Unit of Shimmer3.
Quadriceps thickness | 15 minutes
  Muscular thickness will be analysed using the B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan).
Quadriceps muscle echo-intensity | 15 minutes
  Muscle echo-intensity will be analysed using the B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan).
Mortality | until the end of the study
  examining death rates and risk measures like standardized mortality ratios (SMRs)

CONTACTS AND LOCATIONS:
Locations (1):
- School Medicine University of Malaga, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuentes-Abolafio IJ, Ricci M, Bernal-Lopez MR, Gomez-Huelgas R, Cuesta-Vargas AI, Perez-Belmonte LM. Relationship between quadriceps femoris echotexture biomarkers and muscle strength and physical function in older adults with heart failure with preserved ejection fraction. Exp Gerontol. 2024 Jun 1;190:112412. doi: 10.1016/j.exger.2024.112412. Epub 2024 Apr 6. PMID 38570057
- [Derived] Fuentes-Abolafio IJ, Trinidad-Fernandez M, Ricci M, Roldan-Jimenez C, Gomez-Huelgas R, Arjona-Caballero JM, Escriche-Escuder A, Bernal-Lopez MR, Perez-Belmonte LM, Cuesta-Vargas AI. Kinematic parameters related to functional capacity, fatigue, and breathlessness during the 6-min walk test in older adults with heart failure with preserved ejection fraction. Eur J Cardiovasc Nurs. 2024 Jan 12;23(1):69-80. doi: 10.1093/eurjcn/zvad027. PMID 36808232
- [Derived] Fuentes-Abolafio IJ, Bernal-Lopez MR, Gomez-Huelgas R, Ricci M, Cuesta-Vargas AI, Perez-Belmonte LM. Relationship between quadriceps femoris muscle architecture and muscle strength and physical function in older adults with heart failure with preserved ejection fraction. Sci Rep. 2022 Dec 15;12(1):21660. doi: 10.1038/s41598-022-26064-7. PMID 36522418
- [Derived] Fuentes-Abolafio IJ, Ricci M, Bernal-Lopez MR, Gomez-Huelgas R, Cuesta-Vargas AI, Perez-Belmonte LM. Biomarkers and the quadriceps femoris muscle architecture assessed by ultrasound in older adults with heart failure with preserved ejection fraction: a cross-sectional study. Aging Clin Exp Res. 2022 Oct;34(10):2493-2504. doi: 10.1007/s40520-022-02189-7. Epub 2022 Aug 8. PMID 35939260